CLINICAL TRIAL: NCT01537627
Title: Effects of a Long-term Physical Training Program on Pulmonary and Systemic Aspects in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Long-term Physical Training in Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Fabio Pitta, PhD, PhD, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LFIP-001-NAH-1
Record Dates: First submitted 2012-02-14; First posted 2012-02-23 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Motor activity; Exercise; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-intensity training (LT) (Active Comparator)
  Interventions: Other: Physical training
- High-intensity training (HT) (Active Comparator)
  Interventions: Other: Physical training

INTERVENTIONS:
Other: Physical training — Aerobic exercises (treadmill and cycloergometer): Initially, the intensity is targeted at 60% of maximal capacity and it increases weekly until 110% of maximal capacity. Exercises duration: at least, 20 minutes.
  Resistive exercises (multi gym station; muscle groups: biceps, triceps and quadriceps): Initially, the intensity is targeted at 70% of one maximum repetition (1RM) and it increases weekly until 121% of 1RM. Exercises duration: 3 sets of 8 repetitions. Both exercise training are performed 3 times per week during 6 months.
  Arms: High-intensity training (HT)
Other: Physical training — Callisthenic and breathing exercises are performed during 1 hour, 3 times per week during 6 months. The exercises are divided in 7 different sets and the degree of difficulty of the exercises progresses according to the set.
  Arms: Low-intensity training (LT)

SUMMARY:
Several impairing factors contribute to physical limitation in chronic obstructive pulmonary disease (COPD) as deconditioning, muscle dysfunction and physical inactivity. The available literature clearly indicates that these therapeutic targets benefit from exercise training in patients with COPD and, currently, the key point is not whether patients should or not exercise, but which is the specific contribution of each exercise modality to this population. About this topic, the characteristics of a physical training program to be offered to patients have been a point discussed among researchers in this field, although recently the high-intensity training has been recognized as superior in comparison to the low-intensity training. Literature also indicates that, in order to change the sedentary lifestyle of patients with COPD, long-term training programs are indicated. However, a doubt still remains: if long-term programs are one of the key points to reduce physical inactivity, it is not yet clear whether it is necessary to include high-intensity exercises in that long-term program. If the duration is the only factor influencing the outcomes of the program, thus the intensity of training could be reduced, increasing the adherence of patients to the protocol. Based on this hypothesis, the aim of this study is to compare the effects of two physical training protocols in a long-term rehabilitation program (6 months) in patients with COPD: a high-intensity protocol (based on endurance and resistive training) and a low-intensity protocol (based on callisthenic and breathing exercises training). It is expected that the results of this study contribute to the scientific literature by demonstrating whether low- and high-intensity training contribute equally to change the sedentary lifestyle of patients after a long-term exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Chronic obstructive pulmonary disease (COPD) diagnosis according to Global Initiative for Chronic Obstructive Lung Disease(GOLD)criteria
* Clinical stability (i.e. absence of acute exacerbation in the last 3 months)
* Absence of any unstable/severe cardiac,osteoarticular or neuromuscular disorders which could limit physical activities in daily life
* Non participation in pulmonary rehabilitation in the last year

Exclusion Criteria:

* Being unable to attend the outpatient clinic three times per week
* Inability to understand or cooperate with the assessment methods

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2009-11; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Physical activity in daily life | Up to 4 years
  Main variable: time spent in physical activities of at least moderate intensity (min/day)

SECONDARY OUTCOMES:
Functional exercise capacity | Up to 4 years
  6-minute walking test
Maximal exercise capacity | Up to 4 years
  Incremental Shuttle Walking Test
Peripheral muscle force | Up to 4 years
  1-repetitium maximum and peak quadriceps torque
Respiratory muscle force | Up to 4 years
  Maximal inspiratory and expiratory pressures
Body composition | Up to 4 years
  Electrical Bioimpedance
Health-related quality of life | Up to 4 years
  Chronic Respiratory Disease Questionnaire (CRDQ)
Functional status | Up to 4 years
  London Chest Activity of Daily Living scale (LCADL)
Dyspnea sensation | Up to 4 years
  Borg scale
Lung function | Up to 4 years
  Post-bronchodilator simple spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Pitta, PhD, Study Chair — Laboratory of Research in Respiratory Physiotherapy, State University of Londrina, Brazil; Nidia A. Hernandes, MSc, Study Director — Laboratory of Research in Respiratory Physiotherapy, State University of Londrina, Brazil; Thaís Sant´Anna, PT, Principal Investigator — Laboratory of Research in Respiratory Physiotherapy, State University of Londrina, Brazil; Karina C. Furlanetto, PT, Principal Investigator — Laboratory of Research in Respiratory Physiotherapy, State University of Londrina, Brazil; Leila Donária, PT, Principal Investigator — Laboratory of Research in Respiratory Physiotherapy, State University of Londrina, Brazil
Locations (1):
- Hospital Universitário Norte do Paraná (University Hospital Regional North of Parana), Londrina, Paraná, Brazil